CLINICAL TRIAL: NCT06981312
Title: Internet-Delivered Acceptance and Commitment Therapy for Chronic Pain in Adolescents: A Randomized Controlled Trial.
Brief Title: Internet-Delivered Psychological Treatments for Chronic Pain in Adolescents: ACT and Pain Education.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); Forskningsrådet för hälsa, arbetsliv och välfärd (FORTE) (Unknown)
Responsible Party: Principal Investigator, Charlotte S Gentili, Principal Investigator, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K 2025-3096; 2024-01359 (Other Grant/Funding Number: FORTE: Forskningsrådet för hälsa, arbetsliv och välfärd)
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Nociplastic Pain; Pain Management; Acceptance and Commitment Therapy; Cognitive Behavior Therapy
Keywords: Pain Science Education; Pain Education; Chronic Pain; Nociplastic Pain; Pain Management; Acceptance and Commitment Therapy; Cognitive Behavior Therapy; Adolescent; Parent-Child Relations; Psychological Flexibility; iCBT; Telemedicine
MeSH Terms: conditions — Chronic Pain; Nociplastic Pain; Agnosia | interventions — Acceptance and Commitment Therapy; Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure enhanced Acceptance and Commitment Therapy (Experimental): The treatment protocol to be evaluated focuses on reducing the perceived threat value of pain through pain education, breaking avoidance behaviors through exposure, and increasing the adolescent's psychological flexibility, which are assumed to lead to improvements in function and quality of life. The treatment lasts for nine weeks, during which participants, by accessing information and working with structured exercises, acquire the content of the treatment. The treatment is primarily text-based but also includes images, videos, and audio files. The treatment is provided through the an online platform. Communication with the therapist occurs at least once a week.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Pain Science Education (Active Comparator): This group undergoes the same pain education as the experimental group but with a more comprehensive educational material. The pain education is based on the PSE curriculum. Pain education is relevant as an active control condition, as it is recommended for all patients with at least moderate chronic pain symptoms according to the national care program.
  Interventions: Behavioral: Pain Science Education
- Wait list control (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Participants receive a 9-week internet-delivered intervention: 2 weeks of Pain Neuroscience Education (PNE) based on the PSE curriculum, followed by 7 weeks of Acceptance and Commitment Therapy (ACT) targeting psychological flexibility. In addition to value-oriented behavioral activation, the ACT content includes classical exposure. The treatment is mainly text-based, supported by multimedia content, and delivered on a secure digital platform. Communication with a clinician occurs at least weekly. Parents receive a parallel program based on PSE, ACT, and behavioral principles to support flexible and effective parenting.
  Other Names: Pain education; Exposure therapy
  Arms: Exposure enhanced Acceptance and Commitment Therapy
Behavioral: Pain Science Education — Participants receive 9 weeks of internet-delivered Pain Science Education (PSE), based on the PSE curriculum but with more detailed content, including extended examples, reflection exercises, and behavioral experiments. The aim is to reduce the threat value of pain by promoting a reconceptualization of pain. Parents receive a parallel program with tailored content. The intervention is text-based with multimedia components and delivered via a secure platform. Clinician support is provided asynchronously at least once weekly.
  Arms: Pain Science Education

SUMMARY:
One in four children in Sweden experiences chronic pain. For many, the pain is temporary, but for about 5% it significantly affects daily life, leading to sleep problems, school absence, and reduced physical activity. Youth with chronic pain report lower life satisfaction and overall health compared to their peers. In most cases, there is no underlying disease or injury, suggesting that chronic pain is a condition in itself, driven by dysregulation in the pain system and influenced by biological, psychological, and social factors.

National guidelines in Sweden recommend cognitive behavioral therapy (CBT) and Acceptance and Commitment Therapy (ACT) for children and adolescents with chronic pain and substantial functional limitations. However, more high-quality randomized controlled trials (RCTs) are needed to strengthen the evidence base for these treatments.

The investigators' clinic has developed and evaluated ACT-based treatments for pediatric chronic pain over the past two decades. The protocol has now been adapted into an internet-delivered version to increase accessibility. In a preliminary feasibility study, the investigators observed promising effects on pain interference, though some usability issues have since been addressed.

The treatment is grounded in the fear-avoidance model, which explains how avoidance of pain-related activities can worsen disability over time. In ACT, such avoidance is seen as driven by unwanted thoughts, emotions, and bodily sensations. The aim of treatment is to help young people relate more flexibly to pain and fear and to move toward personally meaningful goals - a skill referred to as psychological flexibility. Exposure is a core component of ACT, encouraging patients to engage with avoided thoughts, feelings, and activities in order to reduce avoidance and improve functioning.

In addition to treating the young person, the study also targets parental behaviors. Parents often respond to their child's pain by increasing protection and monitoring, which is natural but can sometimes contribute to further avoidance and reduced independence in the child. ACT-based parent support is designed to help caregivers support their child more effectively.

In this randomized trial, internet-delivered ACT will be compared to two control conditions: (1) an active comparator involving online pain education, and (2) a passive control group on a wait list. The pain education intervention is based on Pain Science Education (PSE), which aims to shift how individuals understand their pain - from seeing it as a sign of injury to recognizing it as a false alarm in the nervous system. PSE has shown promising effects in adults, but research in youth is still limited, and no RCTs have yet been published.

The study responds to the need for well-designed digital interventions that reach more young people, evaluate treatment components more clearly, and include comparison groups that also receive digital interventions. The goal of the study is to further improve treatment effects by (1) emphasizing exposure strategies to reduce avoidance, (2) expanding pain education to enhance treatment understanding, and (3) refining parent support to better help families manage chronic pain over the long term.

The project aims to increase knowledge about the effects of psychological treatments - in this case delivered online - for adolescents with chronic pain. As previous studies have highlighted the promise of exposure-based strategies and digital accessibility, the study aims to evaluate the effect of a treatment that combines and optimizes both. The study also aims to better understand the specific impact of pain education as a stand-alone intervention, as this is a growing research field with limited studies in youth. Regarding the parent support component of ACT, the study will evaluate whether changes in parental behaviors related to their child's pain are associated with reduced parenting stress and improved functioning and quality of life in the adolescents. In addition to evaluating treatment outcomes, the study aims to explore the underlying processes that may contribute to the effects of ACT and pain education.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13-19 years with chronic pain (duration ≥ 3 months).
* Have undergone a medical examination regarding their pain condition.
* Are not using pain-relieving medication, or have been stable on such medication for at least 2 months, with no planned medication changes.
* Have not undergone ACT or CBT treatment in the past six months.
* Can read and write in Swedish without difficulty.
* Have access to a smartphone/computer with an internet connection and e-ID.
* Have at least one parent or guardian who is willing and able to participate in parallel parent support treatment.

Exclusion Criteria:

* Insufficient understanding of Swedish to complete study-related tasks.
* Adolescents currently undergoing ACT or CBT treatment.
* Adolescents who are using pain-relieving medication or have unstable medication regimes.
* Adolescents without access to a smartphone/computer or e-ID.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain Interference Index | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  Pain Interference Index (PII) is a 6-item self-report questionnaire that assesses the extent to which pain interferes with daily functioning in children and adolescents. Each item is rated on an 11-point scale from 0 to 10, where 0 indicates "no interference" and 10 indicates "complete interference." The total score is the mean of the six items, resulting in a score range from 0 (no interference from pain) to 10 (maximum interference). Higher scores indicate greater interference due to pain.

SECONDARY OUTCOMES:
Psychological Inflexibility in Pain Scale-Avoidance (PIPS-A) | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  The Avoidance subscale of the Psychological Inflexibility in Pain Scale - Adolescent version (PIPS-A) consists of 8 items rated on a scale from 1 (never true) to 7 (always true). Higher scores indicate greater psychological inflexibility through avoidance of pain-related thoughts, feelings, and activities.
KIDSCREEN-10 | Collected at baseline and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  The KIDSCREEN-10 Index is a 10-item measure of health-related quality of life in children and adolescents, with each item rated on a 5-point Likert scale. Raw scores are transformed into T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate better health-related quality of life.
Revised-Childrens Anxiety and Depression Scale 25 (RCADS-25) | Collected at baseline and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  The RCADS-25 is a 25-item self-report scale assessing symptoms of anxiety and depression in children and adolescents. Each item is rated on a 4-point scale from 0 (never) to 3 (always), resulting in a total score ranging from 0 to 75. Higher scores indicate more severe symptoms of anxiety and depression.
Fear of Pain Questionnaire - Child - Short Form (FOPQ-C-SF) | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  The FOPQ-C-SF is a 10-item self-report scale measuring pain-related fear and avoidance in children and adolescents. Each item is rated on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree), yielding a total score ranging from 0 to 40. Higher scores reflect greater fear of pain and avoidance behavior.
Numeric Rating Scale (NRS) - Pain Intensity | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  Pain intensity is assessed using an 11-point Numeric Rating Scale (NRS), where 0 represents 'no pain' and 10 represents 'worst imaginable pain.' Higher scores indicate higher pain intensity.
Numeric Rating Scale (NRS) - Pain Interference | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  Pain interference is assessed using an 11-point Numeric Rating Scale (NRS), where 0 represents 'no interference with daily life' and 10 represents 'completely interferes with daily life.' Higher scores indicate greater interference due to pain.
Pain Reactivity Scale for Parents (PRS-P) | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  The PRS-P consists of 6 items rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 6 to 30, with higher scores indicating greater parental emotional reactivity in response to their child's pain.
School Absence (Parent-Reported) | Collected at baseline and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  Parents report the number of school days missed by their child in the past month due to pain, categorized into intervals: 0-10%, 11-20%, 21-30%, 31-40%, 41-50%, 51-60%, 61-70%, 71-80%, 81-90%, 91-100% of total school days missed.
The Parent Psychological Flexibility Questionnaire (PPFQ-10) | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  A 10-item questionnaire assessing the psychological flexibility of parents in relation to their child's pain. Each item is rated on a 7-point Likert scale, ranging from 1 ("strongly disagree") to 7 ("strongly agree"). Higher scores indicate greater psychological flexibility. The total score can range from 10 to 70, with higher scores reflecting better psychological flexibility in managing stress and responding flexibly to their child's pain-related challenges.
Adult Responses to Children's Symptoms - Protect and Monitor - Youth (ARCS) | Collected at baseline, periprocedural, and directly after completion of the treatment/control condition, as well as at follow-up 3 weeks, 6 months, and 12 months after the end of active treatment.
  This scale assesses the degree to which parents or caregivers respond to their child's pain symptoms with protective and monitoring behaviors. It is typically rated on a Likert scale, where higher scores indicate a higher frequency or intensity of protective and monitoring responses. The total score can vary based on the number of items, but it typically ranges from 0 to a maximum score (for example, 0-24, depending on the number of items on the scale). Higher scores reflect greater protective responses and increased monitoring behavior from the parent or caregiver in reaction to their child's symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Vallentuna, Sweden

IPD SHARING:
Plan to Share IPD: No
Our ethical approval does not allow sharing of individual participant data (IPD).